CLINICAL TRIAL: NCT04637009
Title: A Phase 1 Study of Safety, Pharmacokinetics and Preliminary Activity of TAS1553 in Subjects With Relapsed or Refractory (R/R) Acute Myeloid Leukemia (AML) and Other Myeloid Neoplasms
Brief Title: A Study of TAS1553 in Subjects With Relapsed or Refractory Acute Myeloid Leukemia (AML) and Other Myeloid Neoplasms
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: termination due to portfolio prioritization
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAS1553-01
Record Dates: First submitted 2020-11-15; First posted 2020-11-19 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia; Myeloproliferative Neoplasm; Myelodysplastic/Myeloproliferative Neoplasm
Keywords: MDS/MPN, unclassifiable in chronic phase; Accelerated phase MPN; Chronic neutrophilic leukemia (CNL), accelerated phase; Polycythemia vera (PV), accelerated phase; Primary myelofibrosis (PMF), accelerated phase; Essential thrombocythemia (ET), accelerated phase; Chronic eosinophilic leukemia, not otherwise specified (NOS), accelerated phase; MPN, unclassifiable; MDS/MPN; Chronic myelomonocytic leukemia (CMML); Atypical chronic myeloid leukemia (aCML), BCR-ABL1-negative; MDS/MPN with ring sideroblasts and thrombocytosis (MDS/MPN-RS-T); MDS/MPN, unclassifiable
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myeloproliferative Disorders; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Neutrophilic, Chronic; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Pdgfra-Associated Chronic Eosinophilic Leukemia; Pyloric Stenosis, Hypertrophic; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Thrombocytosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (dose escalation) (Experimental): Oral administration of TAS1553 once daily at specific time points.
  Interventions: Drug: TAS1553
- Part 2 (dose expansion) (Experimental): Oral administration of TAS1553 once daily at specific time points.
  Interventions: Drug: TAS1553

INTERVENTIONS:
Drug: TAS1553 — Form: tablet; Route of Administration: oral

SUMMARY:
This is a Phase 1, 2-part, open-label, multicenter, first-in-human (FIH) study to assess the safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of TAS1553 administered orally to participants ≥18 years of age with relapsed or refractory (R/R) acute myeloid leukemia (AML) or other myeloid neoplasms where approved therapies have failed or for whom known life-prolonging therapies are not available. The AML population includes de novo AML, secondary AML, and myelodysplastic syndrome (MDS)-transformed into AML. Other myeloid neoplasms include accelerated phase myeloproliferative neoplasms (MPN), and chronic or accelerated phase MPN-unclassifiable (MPN-U) and MDS-MPN. Blast crisis phase of MPNs are considered secondary AML and will be included in the AML cohort.

Part 1 is a multicenter, sequential group treatment feasibility study with 1 treatment arm and no masking (dose escalation). Part 2 is a multicenter, two-stage, multiple group, dose confirmation study with 1 treatment arm and no masking (exploratory dose expansion).

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent.
2. Participant must be 18 years of age or older, at the time of signing the informed consent.
3. Life expectancy of at least 12 weeks as assessed by the investigator.
4. Participants with R/R AML or other myeloid neoplasms where approved therapies have failed or for whom known life-prolonging therapies are not available. The AML population includes de novo AML, secondary AML, and MDS transformed into AML. Other myeloid neoplasms include accelerated phase MPN, and chronic or accelerated phase MPN-U and MDS-MPN. Blast crisis phase of MPN, MPN-U, and MDS-MPN are considered secondary AML and will be included in the AML cohort.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Have platelet count ≥10,000/μL (transfusions to achieve this level are allowed).
7. Have adequate renal function as demonstrated by a 24-hour urine measured creatinine clearance ≥60 mL/min.
8. Adequate hepatic function as evidenced by:

   1. aspartate aminotransferase (AST) ≤3× upper limit of normal (ULN)
   2. alanine aminotransferase (ALT) ≤3×ULN
   3. total bilirubin ≤1.5×ULN.
9. Participants must be amenable to serial bone marrow biopsies, peripheral blood sampling, and urine sampling during the study.
10. Women of child-bearing potential (according to recommendations of the Clinical Trial Facilitation Group [CTFG]) must not be pregnant or breastfeeding and must have a negative pregnancy test at screening.

Exclusion Criteria:

1. Participants who have MPN, MPN-U, or MDS/MPN and display hypoplastic bone marrow and would also not ordinarily benefit from cytoreductive therapy such as hydroxyurea (HU).
2. Participants with highly proliferative disease are excluded as follows:

   1. Part 1/AML: white blood cells (WBC) >20,000/μL and >50% blasts in blood. Measures to reduce WBC, such as HU treatment within the last 2 weeks and cytotoxic chemotherapy within the last 4 weeks are not allowed to meet this eligibility criterion.
   2. Part 1/other myeloid neoplasms: WBC >20,000/μL. A short course of HU may be used to meet this eligibility criterion, as long as HU is discontinued 96 hours and any encountered drug-related toxicity must be resolved to Grade ≤1 before the first dose of study treatment.
   3. Part 2/Cohort 1, AML: WBC>20,000/μL and >50% blasts in blood. A short course of HU may be used to meet this eligibility criterion, as long as HU is discontinued 96 hours, and any encountered drug-related toxicity must be resolved to Grade ≤1 before the first dose of study treatment.
   4. Part 2/Cohort 2, other myeloid neoplasms: Specific WBC exclusion criterion not defined. A short course of HU may be used to reduce WBC if judged to be necessary by the investigator, as long as HU is discontinued 96 hours and any encountered drug-related toxicity must be resolved to Grade ≤1 before the first dose of study treatment.
3. Known clinically active central nervous system (CNS) leukemia.
4. Diagnosis of BCR-ABL-positive leukemia, acute promyelocytic leukemia (M3 AML or APML), or juvenile myelomonocytic leukemia (JMML).
5. Second malignancy requiring active systemic therapy, except breast or prostate cancer stable on or responding to endocrine therapy.
6. Ongoing Grade ≥3 Graft Versus Host Disease (GVHD), or any grade GVHD requiring active treatment (for example, calcineurin inhibitors, ≥5mg/day prednisone or other steroid equivalent, or other immunosuppressive agents). (Note: Prednisone at any dose for other indications is allowed).
7. Advanced human immunodeficiency virus (HIV) infection, active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection; Inactive hepatitis carrier status and participants with laboratory evidence of no active replication and participants on antiviral medication(s) who have a viral load below limit of detection will be permitted.
8. Known significant mental illness or other condition such as active alcohol or other substance abuse or addiction that, in the opinion of the investigator, predisposes the participant to high risk of non-compliance with the protocol.
9. Active infection resistant to antibiotics; or non-leukemia-associated pulmonary disease requiring >2 liters per minute oxygen or any other condition that puts the participant at an imminent risk of death.
10. 24-hour urinary protein excretion ≥1g or urinalysis of 2+proteinuria.
11. History of, or at risk for, cardiac disease, as evidenced by any of the following conditions:

    1. Abnormal left ventricular ejection fraction (LVEF; <50%) on echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan at Screening.
    2. Congestive cardiac failure of Class ≥III severity according to New York Heart Association (NYHA) functional classification defined as patients with marked limitation of activity and who are comfortable at rest, while Class IV patients have symptoms of heart failure at rest.
    3. Unstable cardiac disease including unstable angina or hypertension as defined by the need for overnight hospital admission within the last 3 months (90 days).
    4. Ventricular arrhythmias including ventricular bigeminy, clinically significant brady arrhythmias such as sick sinus syndrome, third-degree atrioventricular (AV) block, presence of cardiac pacemaker or defibrillator, or other clinically significant arrhythmias.
    5. Screening 12-lead electrocardiogram (ECG) with measurable QTcF interval of ≥470 msec (Fridericia's formula should be used).
12. Known hypersensitivity to TAS1553 or any of its components.
13. Allogenic hematopoietic stem cell transplantation (HSCT) within 180 days of the first dose of TAS1553, or participants on immunosuppressive therapy post HSCT at the time of screening (calcineurin inhibitors or similar must be discontinued ≥4 weeks prior to the time of study drug initiation).
14. Treated with any systemic anticancer therapy within 2 weeks of the first dose of study treatment. Any encountered treatment-related toxicities (excepting alopecia) must be resolved to Grade 1 or less.
15. Phase 1 Part 1 only: participants who require concomitant use of strong CYP3A4 inducers.
16. Inability to swallow oral medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Safety: Number of participants with treatment-emergent adverse events in Part 1 | Up to 12 months
Safety: Number of participants with dose-limiting toxicities in Part 1 | Up to 12 months
Response rate in Cohort 1 (AML): Number of participants with complete response (CR) + complete response with partial hematological recovery (CRh), and with CR + incomplete blood count recovery (CRi) in Part 2 | Up to 33 months
Response rate in Cohort 2 (other myeloid neoplasms): Number of participants with overall response rate (ORR) of CR + partial response (PR) in Part 2 | Up to 33 months

SECONDARY OUTCOMES:
Pharmacokinetic parameter: Area under the curve (AUC) | At specific timepoints from predose up to Day 8 of Cycle 6 (28 days per cycle)
Pharmacokinetic parameter: Maximum plasma concentration (Cmax) | At specific timepoints from predose up to Day 8 of Cycle 6 (28 days per cycle)
Pharmacokinetic parameter: Minimum plasma concentration (Cmin) | At specific timepoints from predose up to Day 8 of Cycle 6 (28 days per cycle)
Pharmacokinetic parameter: Time to reach maximum plasma concentration (Tmax) | At specific timepoints from predose up to Day 8 of Cycle 6 (28 days per cycle)
Pharmacokinetic parameter: Half-life (t½) | At specific timepoints from predose up to Day 8 of Cycle 6 (28 days per cycle)
Hematological improvement: Number of participants in Cohort 2 (other myeloid neoplasms) with hematological improvement in Part 2 | Up to 33 months
Time to response (TTR): Number of days from the first dose to the first documented evidence of response | Up to 33 months
Duration of response (DOR): Number of days from the start of response until disease progression or relapse | Up to 33 months
Overall survival (OS): Number of days from date of first dose until death due to any cause | Up to 33 months
Safety: Number of participants with treatment-emergent adverse events in Part 2 | Up to 33 months
Pharmacodynamic biomarker: Change from baseline in deoxyadenosine triphosphate (dATP) pool levels in peripheral blood mononuclear cells (PBMCs) | At specific timepoints from predose up to Day 2 of Cycle 2 (28 days per cycle)
Pharmacodynamic biomarker: Change from baseline in phosphorylated checkpoint kinase 1 (pCHK1) levels in bone marrow | At specific timepoints from predose up to Day 2 of Cycle 2 (28 days per cycle)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - University of Alabama - Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - HonorHealth Research Institute, Scottsdale, Arizona
  - University of Southern California Keck School of Medicine, Los Angeles, California
  - Augusta University - Georgia Cancer Center, Augusta, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - Weill Cornell Medicine and New York - Presbyterian Hospital, New York, New York
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Canada (2):
  - University of Alberta Hospital - Hematology Research, Edmonton, Alberta
  - Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No